CLINICAL TRIAL: NCT03480880
Title: Bispectral Index Value Changes During Induction and Surgical Decompression in Head Injury Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIMHANS/DO/103rd IEC/2016
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Traumatic Brain Injury
Keywords: Bispectral Index
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Consciousness Monitors

STUDY DESIGN:
Intervention Model Description: 1. Inj. Thiopentone dose requirement for induction of anaesthesia with and without the use of Bispectral Index guidance.
  2. Observation of Bispectral Index change in intraoperative period.
Who Masked: Participant, Care Provider
Masking Description: 1. Anaesthetic care provider in one arm of first part of study was blinded to intraoperative changes in Bispectral index.
  2. Anaesthetic care provider was blinded to Bispectral Index changes in second part of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BIS (Experimental): Thiopentone dosing during induction of anaesthesia based on guidance of Bispectral Index values.
  Interventions: Device: Bispectral Index
- Group Clinical (No Intervention): Thiopentone dosing during induction of anaesthesia based on clinical guidance targeted to loss of eyelash reflex or loss of response to noxious stimulus.

INTERVENTIONS:
Device: Bispectral Index — Thiopentone was administered in 50 mg boluses during induction of anaesthesia, until reduction of Bispectral Index value to less than 50, and total dose of thiopentone recorded.
  Arms: Group BIS

SUMMARY:
This study was conducted in two parts:

1. This first part was designed to determine thiopentone dose requirement for induction of anaesthesia with and without the use of Bispectral Index monitoring - Participant and Care Provider in appropriate study arm blinded.
2. As a secondary outcome, Bispectral index monitoring was used to observe changes in neuronal function in intraoperative period as well as haemodynamic changes intraoperatively - Participant and Care Provider blinded.

DETAILED DESCRIPTION:
Surgery for traumatic brain injury is an anaesthetic challenge fraught with complications such as brain bulge, excessive bleeding, hypotension etc. As yet there are no anaesthetic regimen guidelines to follow for induction of anaesthesia in neurotrauma surgeries. Although the functional effect of anaesthetic agents on neuronal tissue is known quite well, there is lack of studies documenting the effect of these anaesthetic agents on head injured patients. It is also not known whether the requirement of anaesthetic agent in the same as a non head injured patient. This study was designed to assess the requirement of anaesthetic thiopentone in head injured patients and compare the anaesthetic usage with and without Bispectral index (BIS) monitoring. We also observed the real time change in neuronal function using Bispectral Index monitoring after craniotomy, i.e. effectively decompression and release of intracranial pressure intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Head injury patients coming for surgery

Exclusion Criteria:

* Hypotension/Arrythmias at time of induction
* Extra Dural Hemorrhage
* Extracranial injuries
* Scalp lacerations
* History of Seizures
* No consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Thiopentone requirement | Beginning of anaesthetic induction till End of anaesthetic induction
  Difference of thiopentone requirement with and without use of Bispectral Index guidance during induction of anaesthesia in traumatic brain injury patients.

SECONDARY OUTCOMES:
Intraoperative Bispectral Index changes | Beginning of anaesthetic Induction till patient is shifted to post-anaesthesia care unit.
  Observation of Bispectral Index changes during craniotomy and decompression.
Intraoperative Systolic blood pressure changes | Beginning of anaesthetic Induction till patient is shifted to post-anaesthesia care unit.
  Observation of Systolic blood pressure changes during craniotomy and decompression.
Intraoperative Mean blood pressure changes | Beginning of anaesthetic Induction till patient is shifted to post-anaesthesia care unit.
  Observation of Mean blood pressure changes during craniotomy and decompression.
Intraoperative heart rate changes | Beginning of anaesthetic Induction till patient is shifted to post-anaesthesia care unit.
  Observation of heart rate changes during craniotomy and decompression.

CONTACTS AND LOCATIONS:
Overall Officials: Muthuchellappan Radhakrishnan, MD, DM, Study Chair — National Institute of Mental Health and Neuro Sciences, India

IPD SHARING:
Plan to Share IPD: No